CLINICAL TRIAL: NCT03883035
Title: Utilization of Real-time Automatic Quality-control System in the Detection of Gastric Neoplasms
Brief Title: Quality Control of Esophagogastroduodenoscopy Using Real-time EGD Auxiliary System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yanqing Li (Other)
Responsible Party: Sponsor-Investigator, Yanqing Li, vice president of Qilu Hospital, Shandong University
Organization: Shandong University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2019SDU-QILU-02
Record Dates: First submitted 2019-03-19; First posted 2019-03-20 (Actual); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Esophagogastroduodenoscopy
Keywords: Esophagogastroduodenoscopy; gastric neoplasm; artificial intelligence; quality control
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EAS-aided group (Experimental): esophagogastroduodenoscopy examination with the assistance of automatic quality-control system
  Interventions: Other: automatic quality-control system
- control group (No Intervention): conventional standard esophagogastroduodenoscopy examination without the assistance of automatic quality-control system

INTERVENTIONS:
Other: automatic quality-control system — Automatic quality-control system could real-time measuring endoscopic inspection completeness, detecting gastric neoplasms and evaluating gastric mucosal visibility.
  Arms: EAS-aided group

SUMMARY:
The aim of our study was to develop an automatic quality-control system and assess the performance of this system in quality control of esophagogastroduodenoscopy.

DETAILED DESCRIPTION:
In this study, the researchers firstly developed an automatic quality-control system, name as EAS. Next, the researchers applied the system in a endoscopic center and designed a prospective randomised controlled trial to investigate the performance of the system in quality control of esophagogastroduodenoscopy.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing EGD examination with anaesthesia;
* patients able to give informed consent.

Exclusion Criteria:

* patients with the contraindications to EGD examination;
* patients with a prior EGD examination within 1 year before the trial;
* patients with frankly upper gastrointestinal malignant lesions that were apparent on endoscopy;
* a history of upper gastrointestinal cancers;
* allergic to anaesthetic in previous medical history;
* patients refused to participate in the trial;
* the EGD procedure cannot be completed due to stenosis, obstruction, solid food, or complications of anaesthesia.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1060 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
detection rate of gastric neoplasms | 8 months
  detection rate of gastric neoplasms in different groups

SECONDARY OUTCOMES:
mean number of gastric neoplasms detected | 8 months
  mean number of gastric neoplasms detected per procedure in different groups
mean inspection completeness | 8 months
  inspection completeness per procedure in different groups
mean inspection time | 8 months
  inspection time per procedure in different groups
errors of EAS | 8 months
  errors of EAS in EAS-aided group

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Gastroenterology, Qilu Hospital, Shandong University, Jinan, Shandong, China